CLINICAL TRIAL: NCT05913102
Title: A Prospective, Split-face, Randomized Study of the Poly-D, L Lactic Acid (PDLLA) for Photoaged Skin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jin Cheol Kim (Other)
Responsible Party: Sponsor-Investigator, Jin Cheol Kim, Principal investigator, research assistant professor, Ajou University School of Medicine
Organization: Ajou University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AJOUIRB-INT-2021-630
Record Dates: First submitted 2023-06-10; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Pigmentation; Pigmentation Disorder
MeSH Terms: conditions — Pigmentation Disorders

STUDY DESIGN:
Intervention Model Description: parallel assignment split lesion study
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): administer PDLLA
  Interventions: Drug: PDLLA
- active comparator (Active Comparator): administer saline
  Interventions: Drug: PDLLA

INTERVENTIONS:
Drug: PDLLA — Administer PDLLA/saline every 2 weeks for 2.5 months

SUMMARY:
Juvelook® (VAIM, Korea) is made by dissolving irregular PDLLA particles in a solvent mixture of DMSO (Dimethylsulfoxide) and EC (Ethylene Carbonate) and then injecting them through microneedling to create reticulated foamy microspheres, which are hollow spherical particles. It received CE approval in Europe in 2020 and is widely used domestically as a material for tissue restoration, including skin fillers and collagen stimulators. The spherical shape with internal foam structure of PDLLA exhibits excellent biocompatibility, biodegradability, porosity, and mechanical strength. It allows for the control of particle size and acts as a collagen stimulator while gradually dissolving over time. This stimulates fibroblast cells and promotes skin rejuvenation. In clinical practice, Juvelook® particles are injected to address various concerns such as facial wrinkles, increased elasticity, depressed scars, acne scars, accident scars, under-eye hollows, freckles, whitening effects, and neck wrinkles. Therefore, this study aims to investigate the efficacy of Juvelook® not only in volume augmentation but also in improving photoaged skin.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult women over 30 years old with photoaged skin.
2. Individuals who have a clear understanding of the purpose and content of the study, as well as the potential risks and side effects, and voluntarily sign the informed consent form to participate in the clinical trial.
3. Individuals who are physically healthy and can be tracked and observed throughout the entire study period.

Exclusion Criteria:

1. Individuals who have received anti-aging/whitening treatments (such as laser or chemical peels) on their face within 3 months prior to the start of the study.
2. Individuals who have applied anti-aging/whitening agents to their face within 3 months prior to the start of the study.
3. Pregnant or breastfeeding women.
4. Individuals who are participating in other clinical trials.
5. Individuals who, in the judgment of the researchers, are deemed ineligible to participate in the study.

Min Age: 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-09-28 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
change of lightness value | Chromometer will be taken before treatment and 4,8,12 weeks after last treatment.
  change of lightness value by a chromometer

SECONDARY OUTCOMES:
patinent global assessment for skin condition | Questionnaire will be taken before treatment and 4,8,12 weeks after last treatment.
  patinent global assessment for skin condition by a self-questionnaire
investigator global assessment score for pigmentation | Photos will be taken before each treatment and 4,8,12 weeks after the final treatment.
  investigator global assessment score for pigmentation by clinical photos
Fitzpatrick wrinkle and elastosis scale | Photos will be taken before each treatment and 4,8,12 weeks after the final treatment
  Fitzpatrick wrinkle and elastosis scale by clinical photos

CONTACTS AND LOCATIONS:
Locations (1):
- Ajou University Hospital, Suwon, South Korea

IPD SHARING:
Plan to Share IPD: No